CLINICAL TRIAL: NCT06645769
Title: Na-Phenylbutyrate VAscular Trial
Acronym: NAPVAT
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NAPVAT; R01HL152446 (NIH)
Record Dates: First submitted 2024-10-04; First posted 2024-10-17 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — 4-phenylbutyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NaPB administration (Experimental)
  Interventions: Drug: Sodium Phenylbutyrate
- Placebo control (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sodium Phenylbutyrate — will be compared to placebo
  Arms: NaPB administration
Other: Placebo — will be compared to NaPB
  Arms: Placebo control

SUMMARY:
This study will investigate if the drug sodium phenylbutyrate (NaPB) impacts blood pressure and vascular function in healthy volunteers and in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age and less than 60.
* Healthy subjects will have no history of diabetes or prediabetes.
* Diabetes subjects can be either insulin dependent or not.
* Able to provide written consent and to comply with the procedures of the study protocol.

Exclusion Criteria:

* Age <18 or >60
* Pregnant or lactating women.
* Subjects with hypertension or taking any vasodilatory medications, any steroidal drugs, haloperidol, or valproic acid.
* Patients with congestive heart failure, severe renal insufficiency, hepatic failure, or known sodium retention with oedema.
* Active alcohol or substance abuse.
* Use of tobacco within the previous six months.
* Unble to provide written consent and to comply with the procedures of the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Systemic vascular resistance | from enrollment to the end of participation at 8 weeks
  Arterial hemodynamics and echocardiography to assess systemic vascular resistance, in dynes × sec/cm5.

SECONDARY OUTCOMES:
Plasma BCAAs | from enrollment to the end of participation at 8 weeks
  Plasma branched chain amino acid levels, measured by mass spectrometry (in microMolar)
Flow-mediated dilation (FMD) | from enrollment to the end of participation at 8 weeks
  FMD is a non-invasive test that measures the endothelial function of blood vessels. FMD is measured as a percentage increase in the diameter of an artery during hyperemia (%).
Carotid femoral pulse wave velocity (PWV) | from enrollment to the end of participation at 8 weeks
  Pulse wave velocity (PWV) is the distance a pulse wave travels in a specific arterial segment divided by the time it takes to travel that distance (units: m/sec). PWV is a marker of cardiovascular risk.

OTHER OUTCOMES:
Home ambulatory mean pressure and pulse pressure | from enrollment to the end of participation at 8 weeks
  At home blood pressure cuff used to determine changes in blood pressure with normal activities (mmHg)
Cardiac Ejection Fraction | from enrollment to the end of participation at 8 weeks
  echocardiography will be used to determine ejection fraction (%)

CONTACTS AND LOCATIONS:
Overall Officials: Zoltan Arany, MDPHD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murashige D, Jung JW, Neinast MD, Levin MG, Chu Q, Lambert JP, Garbincius JF, Kim B, Hoshino A, Marti-Pamies I, McDaid KS, Shewale SV, Flam E, Yang S, Roberts E, Li L, Morley MP, Bedi KC Jr, Hyman MC, Frankel DS, Margulies KB, Assoian RK, Elrod JW, Jang C, Rabinowitz JD, Arany Z. Extra-cardiac BCAA catabolism lowers blood pressure and protects from heart failure. Cell Metab. 2022 Nov 1;34(11):1749-1764.e7. doi: 10.1016/j.cmet.2022.09.008. Epub 2022 Oct 11. PMID 36223763
- [Background] Vanweert F, Neinast M, Tapia EE, van de Weijer T, Hoeks J, Schrauwen-Hinderling VB, Blair MC, Bornstein MR, Hesselink MKC, Schrauwen P, Arany Z, Phielix E. A randomized placebo-controlled clinical trial for pharmacological activation of BCAA catabolism in patients with type 2 diabetes. Nat Commun. 2022 Jun 18;13(1):3508. doi: 10.1038/s41467-022-31249-9. PMID 35717342